CLINICAL TRIAL: NCT06234007
Title: Short-course Radiotherapy Followed by Fruquintinib Plus Adebrelimab and CAPOX in the Full Course Neoadjuvant Treatment of Locally Advanced Rectal Cancer: a Multicenter, Single-arm, Open-label Study (UNION PRECISION-I)
Brief Title: Short-course Radiotherapy Followed by Fruquintinib Plus Adebrelimab and CAPOX in the Full Course Neoadjuvant Treatment of Locally Advanced Rectal Cancer: a Multicenter, Single-arm, Open-label Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Tao Zhang, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C128
Record Dates: First submitted 2023-11-13; First posted 2024-01-31 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Neoadjuvant; Fruquintinib; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCRT followed by fruquintinib plus adebrelimab and CAPOX (Experimental)
  Interventions: Drug: Fruquintinib, Adebrelimab, Oxaliplatin, Capecitabine

INTERVENTIONS:
Drug: Fruquintinib, Adebrelimab, Oxaliplatin, Capecitabine — Safety run-in phase: Fruquintinib 4mg/d, oral, once daily, continuous treatment for 2 weeks, 1 week off, q3w, 6 cycles; If the number of patients experiencing dose-limiting toxicity (DLT) was ≤1, the study would continue at that dose level. If the number of patients with DLTs was >1, the dose of fruquintinib was decreased to 3mg/d, qd po, d1-14, q3w, and the dose expansion phase was continued；Adebrelimab 1200mg, d1, IV infusion, q3W, 6 cycles; Capecitabine 1000 mg/m2, twice a day, po, d1-14, followed by 7 days of rest, q3W, 6 cycles; Oxaliplatin 130 mg/m2, d1, q3W, 6 cycles;
  Dose expansion phase: Fruquintinib RP2D, qd po, d1-14, q3w, 6 cycles; Adebrelimab 1200mg, d1, IV infusion, q3W, 6 cycles; Capecitabine 1000 mg/m2, twice a day, po, d1-14, followed by 7 days of rest, q3W, 6 cycles; Oxaliplatin 130 mg/m2, d1, q3W, 6 cycles;

SUMMARY:
To investigate the efficacy and safety of short-course radiotherapy sequential fruquintinib in combination with adebrelimab and CAPOX (full course neoadjuvant therapy) in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study was a multicenter, single-arm, open-label clinical trial. The study included a screening period (within 21 days after signing the informed consent form to the first treatment), a treatment period (including total neoadjuvant and surgical treatment), and a follow-up period (including safety and survival follow-up).

Total neoadjuvant therapy:

* Short-course radiotherapy followed by 6 cycles of fuquinitinib combined with adbelimumab and CAPOX followed by surgical resection after 1 week of rest;
* A treatment time window of ±3 days was allowed during the study treatment, but within 3 days before each treatment, in addition to the required imaging examinations, participants were required to complete laboratory tests, physical examinations (as needed), ECOG scores and other safety assessments to determine that they could still tolerate the study treatment. The safety of the subjects was continuously assessed during the study.
* Total Mesorectal Excision (TME) is recommended for radical resection of rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent and volunteered to participate in the study;
2. Age 18-75 years old (including the cut-off value), male or female;
3. Locally advanced rectal adenocarcinoma confirmed by histopathology;
4. High risk on pelvic MRI [one of the following criteria] :

   * Clinical tumor (cT) stage cT4a or cT4b (according to the AJCC, 8th edition)
   * Extramural vascular infiltration
   * Clinical lymph node (cN) stage cN2 (according to the AJCC, 8th edition)
   * Involvement of the mesenteric fascia
   * Enlarged lateral lymph nodes
5. The distance between the lower edge of the tumor and the anal edge is ≤10cm;
6. Able to swallow tablets and capsules normally;
7. ECOG PS 0-1
8. Have not received any anti-tumor treatment for rectal cancer, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.
9. Plan to undergo surgery after completion of total neoadjuvant therapy;
10. No surgical contraindications;
11. Normal major organ function, including:

    1. Routine blood test (no blood transfusion and blood products within 14 days prior to the first treatment, no correction with G-CSF and other hematopoietic stimulating factors) :

       * Neutrophil count ≥ 1.5×109/L
       * Platelet count ≥ 100×109/L
       * Hemoglobin ≥ 90 g/L
       * White blood cell count ≥ 3.0×109/L
    2. Blood biochemical tests:

       * Total bilirubin ≤ 1.5×ULN (Gilbert's syndrome subjects, ≤3×ULN; Tumor liver metastasis, total bilirubin ≤3×ULN)
       * ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN (≤5×ULN for patients with liver metastases)
       * Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 50 mL/min (Cocheroft-Gault formula, see Annex 2)
    3. Coagulation function:

       * International Normalized ratio (INR) ≤ 1.5×ULN
       * Activated partial thromboplastin time (APTT) ≤ 1.5×ULN
       * Prothrombin time (PT) ≤1.5×ULN
    4. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%
12. Female subjects of childbearing potential were required to have a negative serum pregnancy test within 14 days before starting the trial drug and to have used an effective contraceptive method (e.g., an intrauterine device, contraceptive pill, or condom) during the trial and for at least 6 months after the last dose; Male participants whose partner is a woman of childbearing potential should use effective contraception during the trial and for 6 months after the last dose;

Exclusion Criteria:

1. Previous allergic history to any anti-angiogenesis targeted drug, any component of monoclonal antibody, capecitabine, oxaliplatin, or other platinum drugs;
2. Have received or are receiving any of the following:

   * being treated with an immunosuppressive drug, or systemic hormone, for immunosuppression within 2 weeks before the first dose of the study drug (dose> 10mg/ day prednisone or equivalent); Inhaled or topical steroid use and dosage are allowed in the absence of active autoimmune disease; Prednisone 10mg/ day or equivalent dose of adrenocortical hormone replacement;
   * received live attenuated vaccine within 4 weeks before the first dose of study drug;
   * major surgery or severe trauma within 4 weeks before the first dose of study drug;
3. Have any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered after hormone replacement therapy); Patients with psoriasis or complete remission of childhood asthma/allergies without any intervention in adulthood were considered for inclusion, but patients requiring medical intervention with bronchodilators were not included.
4. A history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation or allogeneic bone marrow transplantation;
5. The presence of uncontrolled cardiac symptoms or diseases, including but not limited to: (1) heart failure above NYHA class II, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias without or poorly controlled after clinical intervention; (5) patients with hypertension that is not well controlled with a single antihypertensive drug (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100mmHg), or patients using two or more antihypertensive drugs to control blood pressure; (6) New York Heart Association (NYHA) functional class > Grade II or left ventricular ejection fraction (LVEF) < 50%;
6. Severe infection (CTCAE > 2) occurred within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications; Prophylactic antibiotics were excluded if there was active pulmonary inflammation on baseline chest imaging, if there were signs and symptoms of infection within 14 days before the first dose of study drug, or if oral or intravenous antibiotics were required;
7. Patients with active pulmonary tuberculosis infection detected by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
8. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive, and HCV RNA above the detection limit of the analytical method);
9. The patient had a second primary malignancy;
10. Pregnant or lactating women;
11. History of arterial/venous thrombosis events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
12. Persons with a history of psychotropic drug abuse and inability to quit or with mental disorders;
13. Patients with any constitutional sign or history of bleeding regardless of severity;
14. Patients with high risk of bleeding, such as active bleeding or bleeding tendency;
15. Urine routine test showed urine protein ≥++, and confirmed 24-hour urine protein quantitation > 1.0 g;
16. According to the investigator's judgment, there are other factors that may lead to the forced termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, alcohol abuse, drug abuse, family or social factors, and factors that may affect the safety or compliance of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pathology complete response(pCR) | up to 6 months
  The proportion of subjects with no residual viable tumor cells(ypT0N0) in the primary tumor and lymph nodes, also defined as the proportion of subjects with grade 0 in the AJCC Tumor Regression Grading (TRG) scoring system(version 8.0).

SECONDARY OUTCOMES:
3-year Event-Free Survival(EFS) rate | up to 36 months
  The percentage of patients without disease recurrence or progression or death due to any cause after 3-year follow-up
Overall Survival(OS) | up to 36 months
  The time from the date of randomization to the death caused by any cause
R0 resection rate | up to 6 months
  The rate of negative margin microscopically
Adverse events (AEs) | up to 36 months
  Adverse events (AEs) were graded according to the NCI CTCAE version 5·0

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; KaiXiong Tao, Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No